CLINICAL TRIAL: NCT06201273
Title: Effects of Two Modalities of Physical Exercise on Physiological Adaptation Capacity, Metabolic Flexibility, and Non-oncological Chronic Pain in Patients Living With Cardiovascular Risk Factors
Brief Title: Physical Exercise on Physiological Adaptation Capacity and Chronic Pain in Individuals With Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, Johnattan Cano Montoya, Academic Researcher, Universidad San Sebastián
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 1662023
Record Dates: First submitted 2023-12-22; First posted 2024-01-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cardiometabolic Risk Factors
Keywords: Exercise; High-Intensity Interval Training; Resistance Training; Interindividual Variability; Intraindividual Variability; Physiological Adaptation; Cardiometabolic Risk Factors; Pain; Chronic Pain; Musculoskeletal Pain; Pain Threshold; Pain Perception; Exercise-Induced Hypoalgesia; Metabolic Flexibility; Indirect Calorimetry; Body Composition; Cardiorespiratory Fitness; Muscle Strength
MeSH Terms: conditions — Motor Activity; Pain; Chronic Pain; Musculoskeletal Pain | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The concealment of allocation will be conducted by a researcher not involved in the clinical procedures of the intervention using the method of opaque, sealed, and consecutively numbered envelopes. The random sequence and allocation concealment allow for the control of selection bias.
  For enhanced bias control, the data analysis will be performed by a researcher blinded to the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Intensity Interval Training (Experimental): This High-Intensity Interval Training (HIIT) program, structured to span 12 weeks, incorporates three sessions per week. Each session comprises 8 to 10 exercise intervals on a cycle ergometer. During these intervals, participants are required to reach an intensity level between 8 and 10 points, based on the modified Borg scale, which ranges from 1 to 10 points. A typical interval involves 1 minute of intensive pedaling, followed by a 2-minute rest period without any activity. To facilitate progressive development, the resistance of the cycle ergometer will be adjusted biweekly to increase the pedaling challenge. Despite these adjustments, participants should consistently maintain their effort intensity within the 8 to 10 point range on the modified Borg scale for each interval.
  Interventions: Behavioral: High-Intensity Interval Training
- Resistance Training (Experimental): This training protocol, spanning a duration of 12 weeks, consists of three weekly sessions. In each session, participants will engage in Elastic Resistance Exercises (ERE) using Theraband elastic bands (CLX). The focus will be on both concentric and eccentric contractions, maintaining an intensity level of 8 to 10 as per the Resistance Exercise Scale (OMNI-RES). Each exercise will be conducted for 1 minute, followed by a 2-minute rest period. Each exercise will be repeated three times within the session.
  The specific exercises include bicep curls, seated horizontal rows, and wide squats. To ensure proper progression and adaptation, the exercise load will be adjusted biweekly. This adjustment will be based on the physiological adaptations of the subjects to the training, aiming to recalibrate the loads to new resistance thresholds and maintain a consistent intensity of 8 to 10 on the OMNI-RES scale for each exercise.
  Interventions: Behavioral: Resistance Training
- Control (No Intervention): Participants in the control group will be instructed to maintain their current lifestyle and exercise habits throughout the duration of the study. This includes adhering to their prescribed medication regimen as usual.

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — This High-Intensity Interval Training (HIIT) program, structured to span 12 weeks, incorporates three sessions per week. Each session comprises 8 to 10 exercise intervals on a cycle ergometer. During these intervals, participants are required to reach an intensity level between 8 and 10 points, based on the modified Borg scale, which ranges from 1 to 10 points. A typical interval involves 1 minute of intensive pedaling, followed by a 2-minute rest period without any activity. To facilitate progressive development, the resistance of the cycle ergometer will be adjusted biweekly to increase the pedaling challenge. Despite these adjustments, participants should consistently maintain their effort intensity within the 8 to 10 point range on the modified Borg scale for each interval.
  Arms: High-Intensity Interval Training
Behavioral: Resistance Training — This training protocol, spanning a duration of 12 weeks, consists of three weekly sessions. In each session, participants will engage in Elastic Resistance Exercises (ERE) using Theraband CLX elastic bands. The focus will be on both concentric and eccentric contractions, maintaining an intensity level of 8 to 10 as per the OMNI-RES scale. Each exercise will be conducted for 1 minute, followed by a 2-minute rest period. Each exercise will be repeated three times within the session.
  The specific exercises include bicep curls, seated horizontal rows, and wide squats. To ensure proper progression and adaptation, the exercise load will be adjusted biweekly. This adjustment will be based on the physiological adaptations of the subjects to the training, aiming to recalibrate the loads to new resistance thresholds and maintain a consistent intensity of 8 to 10 on the OMNI-RES scale for each exercise.
  Arms: Resistance Training

SUMMARY:
This research focuses on studying the effects of a 12-week exercise program on the health of individuals at risk of heart disease. The program includes High-Intensity Interval Training (HIIT) and Muscle Endurance Resistance Exercise (ERE). The researchers aim to observe the impact of these exercises on physiological adaptability, physical capacity, cardiovascular risk factors, metabolism, body composition, and chronic pain.

The participants will be inactive adults with a Body Mass Index (BMI) between 25 and 39.9, who are enrolled in a cardiovascular health program. Individuals with certain serious conditions, such as bone or heart problems, pulmonary diseases, cancer, or those who do not adequately understand instructions or Spanish, are ineligible to participate.

Patients will be selected by the program team and divided into three groups: one will perform HIIT, another will engage in ERE, and a control group will continue their usual treatment. Participants will be assessed at different times: before starting, at 4 weeks, at 8 weeks, and at the end of the program. Various health aspects will be measured, including physical activity, quality of life, physical capacity, cardiovascular risk factors, metabolism, body composition, and pain level.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive: Not engaging in 300 minutes of moderate or 150 minutes of vigorous physical activity per week, measured with the IPAQ questionnaire.
* BMI between 25 and 39.9 kg/m².
* Belonging to the cardiovascular health program of External Family Health Center Valdivia.
* Presenting or not presenting chronic non-cancerous pain.

Exclusion Criteria:

* Bone disease.
* Ischemic disease or arrhythmia.
* Chronic obstructive pulmonary disease (COPD) or asthma.
* Uncontrolled chronic diseases.
* Individuals unable to understand instructions.
* Individuals who do not speak Spanish.
* History of previous oncological disease or under investigation for suspected neoplastic disease in any part of the body.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Systolic and Diastolic Blood Pressure | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Pressure in the arteries during and between heartbeats. (mmHg)
Heart Rate | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Number of heartbeats per minute. (bpm)
Body Composition | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Percentage of Fat and Lean Mass: Proportion of fat and lean mass in the body. (%)
Metabolic Flexibility | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Indirect Calorimetry: Measurement of energy expenditure and substrates balance. (kcal)
Pain Intensity: | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  The Chronic Pain Grade Scale is a self-report instrument assessing the intensity and disability associated with chronic pain. It comprises 8 items, 7 of which are in an 11-point Likert format, totaling a range from 0 to 70 points. The final score is derived from summing items 2 to 8.
  Items 2, 3, and 4 address pain intensity, while items 5, 6, 7, and 8 pertain to disability related to chronic pain.
  Chronic pain grading based on this scale is classified as:
  Grade I (low intensity): considering less than 15 points in pain intensity items and less than 17 points in disability items.
  Grade II (high intensity): 15 points or more in pain intensity items and less than 17 points in disability items.
  Grade III (moderately limiting): 17 to 24 points in disability items.
  Grade IV (severely limiting): 25 to 40 points in disability items.
Pressure Pain Threshold (PPT): | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Pressure Algometer Measurement: Minimum amount of pressure that induces pain. (kg)
Pain Characterization: | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  The characterization of chronic pain will be conducted using questions 15 and 16 (based on the neuropathic pain 4 questionnaire) from the 2013 validated Chilean survey of non-oncological chronic pain.
  These questions allow for the categorization of pain as either somatic or neuropathic, as detailed below:
  Somatic Pain: Sharp, widespread (in a nonspecific area), a specific area related to some movement, a squeeze.
  Neuropathic Pain: Burning, cold pain, electric, tingling, prickling, itching, needle sensation, numbness.
Handgrip strength | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Handgrip Dynamometry: Measurement of handgrip strength. (kgf or N)
Cardiorespiratory fitness | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  6-minute walk test: The objective is to assess an individual's functional capacity and cardiorespiratory endurance. The primary measurement unit is the distance covered in meters during the 6 minutes
Fasting Glucose | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Blood glucose level after a fasting period. (mg/dL)
Glycated Hemoglobin (HbA1c): | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Percentage of glucose-bound hemoglobin in the blood. (%)
Lipid Profile | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Set of tests to measure cholesterol and triglycerides. (mg/dL)

SECONDARY OUTCOMES:
Sociodemographic and Medical Background | Pre-Intervention: Initial assessment before the training
  * Gender: Biological classification of the individual. (No unit of measure)
  * Age: Number of complete years since birth. (Years)
  * Ancestry: Ethnic or racial origin of the individual. (No unit of measure)
  * Education Level: Highest level of education achieved. (No unit of measure)
  * Duration in Cardiovascular Health Program: Length of participation in the program. (Months or Years)
  * Morbid Background: History of previous diseases and medical conditions. (No unit of measure)
  * Medications and Dosage: Description of used medications and their dosages. (mg/day or as prescribed)
  * Duration of Medication Use: Length of time medications have been used. (Months or Years)
Physical Activity Level | Pre-Intervention: Initial assessment before the training.
  The International Physical Activity Questionnaire (IPAQ) is a recognized instrument for assessing physical activity in adults. This survey outlines the frequency (measured in days per week) and duration (hours and minutes per day) of physical activities categorized into four intensity levels: sedentary, walking, moderate physical activity, and vigorous physical activity.
  For each intensity level, the units of measurement are expressed in days per week and hours or minutes per day, with specific Metabolic Equivalent Task (METs) values assigned to each activity (Walking: 3.3 METs, Moderate Physical Activity: 4 METs, Vigorous Physical Activity: 8 METs). The responses can be converted into MET-minutes/week, enabling a quantitative and consistent comparison of total physical activity, encompassing various types and intensities.
Health-related quality of life | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  The (Short Form Health Survey - 36 is a questionnaire designed to measure health-related quality of life. It consists of 36 items covering eight health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Each domain is scored separately, and the scores are transformed into a 0 to 100 scale, where a higher score indicates better quality of life or less impact of the illness in that dimension.
Height | Pre-Intervention: Initial assessment before the training.
  Individual's height. (cm)
Weight | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Total body mass. (kg)
Body Mass Index | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  The Body Mass Index (BMI) is a metric used to assess the relationship between an individual's weight and height, thereby estimating their weight category, which can range from underweight to obesity. It is calculated by dividing a person's weight in kilograms by the square of their height in meters.
  The formula is: BMI = weight (kg) / [height (m)]^2
  The unit of measurement for BMI is kg/m² (kilograms per square meter).
Waist Circumference | Pre-Intervention: Initial assessment before the training. Week 4: Mid-program evaluation. Week 8: Eight-week assessment. Post-Intervention (Week 12): Final evaluation after 12 weeks.
  Measurement of the abdominal circumference. (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Johnattan Cano Montoya, Principal Investigator — Universidad San Sebastián
Locations (1):
- Universidad San Sebastián, Valdivia, Los Ríos Region, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cano-Montoya J, Rojas Vargas M, Baez Vargas S, Nunez Vergara C, Martinez Huenchullan S, Gallegos F, Alvarez C, Izquierdo M. Impact of resistance and high-intensity interval training on body composition, physical function, and temporal dynamics of adaptation in older women with impaired cardiometabolic health: a randomized clinical trial. BMC Sports Sci Med Rehabil. 2025 Apr 11;17(1):78. doi: 10.1186/s13102-025-01119-0. PMID 40217506

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT06201273/Prot_SAP_ICF_000.pdf